CLINICAL TRIAL: NCT04112550
Title: Clinical Effectiveness of Pre-operative Methadone in Single Level Lateral Transpsoas Interbody Fusions: A Randomized, Double-blinded, Controlled Trial
Brief Title: Clinical Effectiveness of Pre-operative Methadone in Single Level Lateral Transpsoas Interbody Fusions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, SBarber, Neurosurgery Faculty, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00022567
Record Dates: First submitted 2019-09-27; First posted 2019-10-02 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Degenerative Disc Disease; Spondylolisthesis, Lumbar Region
Keywords: lateral lumbar interbody fusion; minimally invasive spinal surgery
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis | interventions — Methadone; oxycodone-acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Methadone (Active Comparator): This cohort will receive oral methadone 15mg po tablet pre-operatively
  Interventions: Drug: Methadone Hydrochloride
- Oxycodone (Active Comparator): This cohort will receive oxycodone/acetaminophen 10/325 po tablet pre-operatively
  Interventions: Drug: Oxycodone-Acetaminophen

INTERVENTIONS:
Drug: Methadone Hydrochloride — FDA approved medication to treat pain
  Arms: Methadone
Drug: Oxycodone-Acetaminophen — FDA approved medication to treat pain
  Arms: Oxycodone

SUMMARY:
Spinal operations including lumbar fusions for degenerative disorders are becoming more prevalent as the population ages. Inadequate or excessive postoperative analgesia can result in medical comorbidities and prolonged hospital length of stay and patient dissatisfaction.

Existing literature has highlighted the preoperative administration of methadone as a promising adjuvant for post operative pain control. Methadone has the benefit of being long-acting and has more stable serum concentration and a single preoperative dose may have significant benefits post operatively.

Here the investigators propose a prospective parallel-group, randomized, double-blinded study to assess post operative analgesic requirements after preoperative administration of either methadone 15 mg or Oxycodone 10/325. Primary outcome will be total IV and PO narcotic consumption in the post operative course. Secondary outcomes examined will include time to mobility, need for specialist pain management consultation, early readmission (within 2 weeks) for inadequate pain control, and complications associated with administration.

DETAILED DESCRIPTION:
Lumbar spinal fusions are becoming increasingly popular and prevalent in the treatment of a variety of spinal pathologies, but predominantly for degenerative disease which is most prevalent in the obese and or older population. These operations can result in relatively high post operative surgical pain and necessitate significant post operative opioid consumption which can precipitate co-morbid medical conditions such as respiratory depression and failure, pneumonia, gastrointestinal ileus, deep venous thrombosis, and pulmonary embolism. Additionally, these medical comorbidities also represent an increased burden on healthcare expenditure with increased length of hospital stay, inpatient testing and treatment, and need for additional follow up.

The investigators objective is to study the effect of a long term opioid analgesic, methadone, in a uniform population undergoing a single level minimally invasive lumbar fusion. The preoperative single dose administration of methadone has already been shown to be effective in improving post operative pain control in open multi-level spinal fusion patient populations and has become the standard of care in most surgical centers across the country. The long half-life of methadone results in improved steady state pharmacokinetics relative to other traditional opioids and is thought to improve pain control while decreasing consumption. In addition to Mu opioid receptor agonism, Methadone is thought to also have adjunctive analgesic and anti-tolerance effects due to CNS excitatory glutamatergic NMDA receptor antagonism. There are also reports of synergistic effects from serotonin and norepinephrine reuptake inhibition.

The investigators predict that a single preoperative oral methadone administration can result in improved postoperative analgesia with requirement of less IV and PO traditional narcotics within the first 2 weeks post operatively and also will not increase co-morbid risks relative to traditional shorter acting opioid analgesics that are presently given preoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 70
* Will undergo one level minimally invasive lumbar fusion surgery
* Primary symptoms are back and/or leg pain

Exclusion Criteria:

* Preoperative chronic renal insufficiency or failure (defined as a serum creatinine more than 2 mg/dl)
* Significant liver disease (cirrhosis or hepatic failure)
* American Society of Anesthesiologists (ASA) physical status IV or V
* Pulmonary disease necessitating home oxygen therapy
* Patients with acute bronchial asthma or hypercarbia
* Patient who has or is suspected of having a paralytic ileus
* Preoperative use of methadone or hydromorphone
* Known hypersensitivity to methadone
* Known hypersensitivity to oxycodone
* Recent history of opioid or alcohol abuse
* Inability to use a PCA device
* Inability to speak English
* Any patient judged by the anesthesia care team to potentially require prolonged postoperative intubation
* Participation in another clinical trial
* Inability of patient to provide study informed consent (including patients who are cognitively impaired)
* Presence of drug interaction between methadone/oxycodone and patient's regular or PRN medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-02-11 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative in-hospital patient's narcotic requirement | Post-operative day 0 to 4
  The total Morphine Milligram Equivalent (MME) for each post-operative day
Improvement in low back pain between the two cohorts as assessed by Oswestry Disbility Index (ODI) | 14 days
  Change in ODI (scale from 0 to 100) from pre-op to post-op (14 days post-op)

CONTACTS AND LOCATIONS:
Overall Officials: Sean M Barber, MD, Principal Investigator — The Methodist Hospital Research Institute

IPD SHARING:
Plan to Share IPD: Undecided
No plans to share IPD at the moment